CLINICAL TRIAL: NCT00480259
Title: Hyperproteic Nutrition; Correlation of BUN to Nitrogen Balance and Associated Infection Rates With Bimodal Protein Administration
Brief Title: Hyperproteic Nutrition:Correlation of BUN to Nitrogen Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25351
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Enteral Feeding
Keywords: blood urea nitrogen; nitrogen balance; nutrition; intensive care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Nutrition (Active Comparator)
  Interventions: Behavioral: hyperproteic nutrition
- Hyperprotein Nutrition (Experimental)
  Interventions: Behavioral: hyperproteic nutrition

INTERVENTIONS:
Behavioral: hyperproteic nutrition

SUMMARY:
This study is designed to determine if the following are true. When protein requirements exceed metabolic requirements, blood urea nitrogen(BUN) levels will rise. Elevated BUN levels in the absence of renal failure, hepatic failure, or GI bleeding, will be correlated with improved nitrogen balance and inversely correlated with infection rates, days of mechanical ventilation, ICU days, and total hospital days.

DETAILED DESCRIPTION:
The purpose of this study is threefold. First, to determine if a correlation exists between BUN and nitrogen balance in the context of hyperproteic nutrition administration. Creatinine clearance will also be followed to determine if there is any harmful effect to the kidney secondary to an elevated BUN. Secondly, to determine if there is a difference in hospital acquired infection rate, ventilator days, ICU days, and hospital stay between the current nutrition standard at Penn State Hershey Medical Center and a hyperproteic nutrition protocol. Thirdly, to determine the accuracy of at least three calculated creatinine clearance formulae when compared to a measured creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

* Greater then or equal to 18 years of age and patient in Intensive Care Unit
* Receiving enteral nutrition, with expected duration of at least 5 days
* Blood urea nitrogen and creatinine clearance are part of routine blood work
* Indwelling urinary catheter in place

Exclusion Criteria:

* Renal or hepatic failure
* Current or history(past 6 mos) of GI bleeding
* Serum creatinine on day of screening of equal to or greater then 1.5 mg/dl
* Creatinine Clearance on day of screening of equal to or less then 30ml/min
* Hypovolemia resulting in increased BUN
* Septic shock
* Blood urea nitrogen on day of screening equal to or greater then 30mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2009-04-21 (Actual); Study Completion 2009-04-21 (Actual)

PRIMARY OUTCOMES:
Increase in BUN | Unable to document -incomplete information and investigator no longer at institution; no records available

SECONDARY OUTCOMES:
Decrease in infection rate, ventilator days, ICU stay and hospital dys | Unable to document -incomplete information and investigator no longer at institution; no records available

CONTACTS AND LOCATIONS:
Overall Officials: John K Stene, MD, Principal Investigator — Penn State University, College of Medicine, Dept of Anesthesiology